CLINICAL TRIAL: NCT06824389
Title: Evaluate the Performance of Large Language Models in Ophthalmologic Patient Consultation: A Randomized Clinical Trial
Brief Title: Evaluate the Performance of Large Language Models in Ophthalmologic Patient Consultation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2025KYPJ004
Record Dates: First submitted 2025-02-05; First posted 2025-02-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Non-emergency Ocular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large language models in consultation (Experimental): After the patient signs the informed consent form, the large language model completes the medical history collection and recommends examinations.
  Interventions: Other: Consultation Model of large language model in Ophthalmology Clinics
- Traditional consultation (No Intervention): After the patient signs the informed consent form, doctor completes the medical history collection and recommends examinations.

INTERVENTIONS:
Other: Consultation Model of large language model in Ophthalmology Clinics — Large language model completes the medical history collection and recommends examinations.
  Arms: Large language models in consultation

SUMMARY:
The intelligent image models lack an understanding of diagnostic and treatment logic, and have not considered textual information such as symptoms and signs. Large language models like ChatGPT, can learn medical knowledge, understand, and generate human natural language, offering new technologies for medical knowledge-based intelligent question answering and the creation of smart medical documents. Therefore, our team plan to verify large language models' feasibility and effectiveness in ophthalmology clinics for medical history collection and examination recommendations during consultations, comparing its performance with traditional methods.

ELIGIBILITY:
Inclusion Criteria:

* No age or gender restrictions for patients.
* Non-emergency ocular diseases including corneal diseases, lens disorders, and vitreoretinal diseases.
* Voluntary participation with signed informed consent.

Exclusion Criteria:

* Top 10 Ocular Emergencies: globe perforation, ocular chemical injury, corneal ulcer perforation, Pseudomonas aeruginosa keratitis, acute angle-closure glaucoma, acute panophthalmitis, central retinal artery occlusion, acute optic neuritis, endophthalmitis, and orbital cellulitis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Medical History Collection Scoring | through study completion, up to 1 week.
  The medical history collection is performed using the standard outpatient medical record form. The scoring criteria are developed collaboratively by clinical doctors from multiple specialties and researchers. Scoring is independently conducted in a blinded manner by higher-level specialists.

SECONDARY OUTCOMES:
Accuracy of Recommended Tests | through study completion, up to 1 week.
  The gold standard for both the experimental and control groups consists of test items independently selected by senior specialists, who are not involved in the study.
Duration of Medical History Collection | through study completion, up to 1 week.
  The experimental group uses the developed system to record the consultation and medical record writing completion times, while the control group records the consultation time through audio recording and the medical record writing completion time through the developed system.
Patient satisfaction | through study completion, up to 1 week.
  Collected through a questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No